CLINICAL TRIAL: NCT01345188
Title: Ranolazine in Ischemic Cardiomyopathy Patients With Persistent Chest Pain or Dyspnea Despite Conventional Therapy: A Cross-Over Study
Brief Title: Ranolazine in Ischemic Cardiomyopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Midwest Cardiovascular Research Foundation (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Dr. Nicolas Shammas, Principal Investigator, MD, Midwest Cardiovascular Research Foundation
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IN-US-259-D032
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Results first posted 2018-09-06 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Cardiomyopathy; Chest Pain; Dyspnea
MeSH Terms: conditions — Cardiomyopathies; Chest Pain; Dyspnea | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine (Active Comparator): 1000 mg Ranexa orally once daily titrated as tolerated after 1 week up to taking 1000 mg twice daily.
  Interventions: Drug: Ranexa
- Placebo (Placebo Comparator): 1000 mg placebo orally once daily titrated as tolerated after 1 week up to taking 1000 mg twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranexa — 1000 mg Ranexa orally once daily titrated as tolerated after 1 week up to taking 1000 mg twice daily.
  Other Names: Ranolazine
  Arms: Ranolazine
Drug: Placebo — 1000 mg placebo orally once daily titrated as tolerated after 1 week up to taking 1000 mg twice daily.
  Arms: Placebo

SUMMARY:
Patients with ischemic cardiomyopathy may continue to experience persistent chest pain and shortness of breath despite conventional medical therapy and/or revascularization. The purpose of this study is to determine the efficacy of taking Ranexa versus placebo in patients with ischemic (due to blockages) cardiomyopathy treated with optimal conventional medical therapy and/or percutaneous revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic cardiomyopathy patients on optimal medical treatment. Optimal medical treatment is defined as the continued symptoms of chest pain or dyspnea despite treatment with 2 antiischemic agents (beta blockers, CCB or nitrates). Unless contraindicated, all cardiomyopathy patients should be treated with a beta blocker and an ACEI/ARB.
2. Anginal chest pain or dyspnea
3. Documentation of non treatable or optimally treated coronary artery disease
4. Ejection Fraction of less than or equal to 40%

Exclusion Criteria:

1. Less than 18 years of age
2. Pregnant or breast feeding
3. Patients with non ischemic cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas W Shammas, MD, Principal Investigator — Midwest Cardiovascular Research Foundation
Locations (1):
- Midwest Cardiovascular Research Foundation, Davenport, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from a cardiovascular clinic in Davenport, Iowa between 5/21/2012 and 11/22/2013
Pre-assignment Details: A total of 36 patients assessed for eligibility. Excluded were 8 patients (did not meet inclusion criteria=4; declined to participate=3;other=1). 28 patients were included in this randomized cross-over study.
Groups:
- Ranolazine, Then Placebo: Patient received Ranolazine to 1,000 mg ranolazine orally twice a day, as tolerated for 6 weeks. After a washout period of 2 weeks, they then received Placebo tablet (matching Ranolazine 1000 mg tablet twice a week) for 6 weeks.
Period: Randomization Ranolazine/Placebo 6 Weeks
Arm/Group | Ranolazine, Then Placebo
Started | 28
Completed | 26
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Crossover Ranolazine/Placebo 6 Weeks
Arm/Group | Ranolazine, Then Placebo
Started | 26
Completed | 25
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes both groups randomized to placebo and ranolazine
Arm/Group | Entire Study Population
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 23
Ejection Fraction [Mean (Standard Deviation); unit: Percentage] | 33.1 (7.6)
Diabetes Mellitus [Number; unit: participants] | 19
Prior myocardial infarction [Number; unit: participants] | 23

OUTCOME MEASURES:

1. Primary Outcome: Anginal Frequency
Description: Anginal frequency as assessed by Seattle Angina Questionnaire. Scoring is done by assessing responses on an ordinal value. Anginal score is scored by the patient by selecting a number from 0 to 100 with low score indicates more anginal frequency. The mean of the the scores of all patients analyzed were compared between placebo and Ranolazine.
Time Frame: 12 weeks
Population: Patients receiving ranolazine for 6 weeks and crossed over to placebo or vice versa. Higher number on the angina scale indicates less angina
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Placebo: Patients that received placebo
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | 86.67 [40 to 100] | 74.44 [10 to 100]
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority or Other; p = 0.058, Paired t test

2. Primary Outcome: Quality of Life Questionnaire
Description: Quality of life as measured by the Seattle Angina Questionnaire as a score ranging from 0 to 100. Higher score indicates better quality of life. The Qaulity of life is scored by the patient. It assesses the perceived satisfaction or dissatisfaction in the major domains of life.
  These include mobility, self-care, Usual activities (leisure, work, family), Pain/Discomfort, and Anxiety.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Ranolazine: Patients that received ranolazine
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | 72.22 [50 to 92] | 66.67 [42 to 92]
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority or Other; p = 0.048, Paired t test

3. Primary Outcome: Dyspnea Assessed by the Rose Dyspnea Questionnaire (RDQ)
Description: RDQ is a four item questionnaire that evaluates a patient's dyspnea with regular activity. Each question answered postiviely is given a score of 1. Total score possible is 4. A higher score indicates worse dyspnea. A difference between the score at end of treatment minus baseline is performed. A negative score indicates improvement. Comparing the difference between the 2 arms (placebo and ranolazine) is performed.
Time Frame: 12 weeks
Population: Patients with dsypnea. The score reflects difference between baseline and following treatment with ranolazine or placebo
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -0.45 [-4 to 2] | -0.34 [-2 to 1]
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority or Other; p > 0.05, Wilcoxon Signed rank

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Ranolazine: patients receiving ranolazine
- Placebo: Patients receiving placebo
Arm/Group | Ranolazine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/24
Other Adverse Events (participants affected / at risk) | 6/24 | 2/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=24) | Placebo (N=24)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) — patient was admitted to the hospital with exacerbation of his heart failure, but this patient also had pneumonia and sepsis.study drug.
stroke (Nervous system disorders) | 1 (1) | 0 (0) — From atrial fibrillation. Unrelated to study medication
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=24) | Placebo (N=24)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) — Intolerance to high dose of medication
diziness (Nervous system disorders) | 3 (3) | 2 (2) — Intolerance to medication
constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No